CLINICAL TRIAL: NCT03319563
Title: High Volume, Multilevel Local Anesthetic-Epinephrine Infiltration in Kyphoscoliosis Surgery: Blood Conservation and Analgesia
Brief Title: Kyphoscoliosis Surgery: Blood Conservation and Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Alaa Mazy Mazy, Associate professor of anesthesia and surgical intensive care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R/17.02.85; PACTR201703002123104 (Registry Identifier: the Pan African Clinical Trial Registry)
Record Dates: First submitted 2017-10-11; First posted 2017-10-24 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Posterior Spine Surgery
MeSH Terms: interventions — Sodium Chloride; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local anesthetic-epinephrine group (Experimental): after general anesthesia, the Infiltration cocktail was done by the surgeon at three levels:
  1. Subcutaneous: before incision at a volume 20 ml/10 cm/side.
  2. Muscular Paravertebral: before opening the thoracolumbar fascia, using the same previous volume.
  3. Neural paravertebral: after exposure of the transverse processes. A volume of 5 ml/per each process of the same cocktail, 1 cm deep to the surface of the corresponding process before pedicular screws fixation after negative blood aspiration.
  Interventions: Drug: Local anesthetic-epinephrine
- saline group (Placebo Comparator): after general anesthesia, the same infiltration volume and technique using normal saline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Local anesthetic-epinephrine — * Bupivacaine 0.5% (Astra Zeneca) 2 mg/Kg.
  * Lidocaine 5 mg/Kg.
  * Epinephrine 5 mcg/ml of the total volume.
  * Add normal saline to a total volume of 100 ml/10 cm of the wound length.
  Other Names: infiltration group
  Arms: local anesthetic-epinephrine group
Drug: Saline — normal saline 100 ml/10 cm of the wound length
  Other Names: control group
  Arms: saline group

SUMMARY:
Since the first spinal fusion by Hibbs 1911, yet anesthesia for correction of scoliosis is challenging due to frequently associated co-morbidities, the extensive nature of surgery and liability for many complications. Among the major concerns for anesthesiologists are the pain and bleeding. Scoliosis correction accounts for massive blood loss that may exceed more than half of blood volume. There are many strategies for blood conservation; however sometimes some of them may not be suitable. For analgesia, the most frequently loco regional analgesic techniques in spine surgery are intrathecal, epidural or local infiltration techniques. infiltration data reviled inconclusive and heterogeneous results. Our purpose is to optimize blood conservation and analgesia through anatomically based modification of the infiltration technique.

DETAILED DESCRIPTION:
The most frequently loco-regional analgesic techniques in scoliosis surgery are intrathecal, epidural, caudal morphine, or local infiltrations techniques including ultrasound guided thoracolumbar interfascial plane block. however these techniques possess some limitations in scoliosis surgery. Local anesthetic infiltration was first applied over 35 years ago in lumbar spine surgery as a reliable technique for pain relief. However meta-analysis of data reviled inconclusive and heterogeneous efficacy results.This conflict arise from the differences in the technique and drugs.There are three levels of infiltration; subcutaneous, muscular and perineural. Its timing either pre-incision or post-surgery. Generally the preemptive and deep infiltration offer better analgesia when compared with post-surgical and superficial forms. Different drugs including local anesthetics, epinephrine and adjuvants can be given as a single injection or infusion. Doses and volumes are also different, usually ranging from 10 to 30 ml at a concentration of 0.25% Bupivacaine. the use of epinephrine helps bleeding control Concomitantly, unlike the other techniques, bupivacaine infiltration was combined at three levels in this study; subcutaneous, muscular and neural paravertebral to provide sensory, motor and sympathetic blockade all together. In addition, this drug combination may help to maintain spinal cord perfusion by avoiding deliberate hypotension. The high volume sufficient for proper tissue infiltration combined at three anatomically guided levels for three types of nerves has not been described so far. This research may benefit all spine surgery patients.

ELIGIBILITY:
Inclusion Criteria:

1. Kyphoscoliosis patients subjected for spinal correction.
2. Age 8-18 years.
3. American Society of Anesthesiologists I-II status.

Exclusion Criteria:

1. Patient or parents refusal.
2. Infection at surgical site.
3. Hypersensitivity to amide local anesthetics.
4. Coagulopathy.
5. Blood diseases as sickle cell anemia, hemophilia, idiopathic thrombocytopenic purpura.
6. Sever cardiac, respiratory, renal or hepatic impairment.
7. Presence of communication barrier.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | Intraoperative
  milliliter
Total Morphine consumption. | during first 24 hours postoperatively.
  milligram

SECONDARY OUTCOMES:
The surgical field visualization for subcutaneous incision | Intraoperative, 10 minutes after skin incision.
  measured by Fromme's operative visibility scale (0-5) ,5: Massive uncontrollable bleeding, Surgery impossible. 4: Heavy but controllable. 3: Moderate bleeding , 2: Moderate bleeding but without interference with accurate dissection. 1: Bleeding, so mild, No suctioning. 0: No bleeding,
The surgical field visualization for muscular dissection | Intraoperative, 30 minutes after the thoracolumbar fascia incision,
  measured by Fromme's operative visibility scale (0-5) ,5: Massive uncontrollable bleeding, Surgery impossible. 4: Heavy but controllable. 3: Moderate bleeding , 2: Moderate bleeding but without interference with accurate dissection. 1: Bleeding, so mild, No suctioning. 0: No bleeding,
The surgical field visualization for nails insertion | Intraoperative, 30 minutes after the first nail insertion.
  measured by Fromme's operative visibility scale (0-5) ,5: Massive uncontrollable bleeding, Surgery impossible. 4: Heavy but controllable. 3: Moderate bleeding , 2: Moderate bleeding but without interference with accurate dissection. 1: Bleeding, so mild, No suctioning. 0: No bleeding,
The surgical field visualization for osteotomy | Intraoperative, 20 minutes after the first osteotomy
  measured by Fromme's operative visibility scale (0-5) ,5: Massive uncontrollable bleeding, Surgery impossible. 4: Heavy but controllable. 3: Moderate bleeding , 2: Moderate bleeding but without interference with accurate dissection. 1: Bleeding, so mild, No suctioning. 0: No bleeding,
The operative duration | Intraoperative
  minutes, from the start of anesthesia induction to extubation times
The number of blood transfusion unites. | intraoperative
  unites of packed red blood cells
Nitroglycerin consumption | Intraoperative
  milligram
Fentanyl consumption | intraoperative
  microgram
Atracurium consumption | intraoperative
  milligram
Propranolol consumption | intraoperative
  milligram
Mean blood pressure (MBP) | basal, 5 minutes after the onsite of infiltration, 3 minutes after the onsite of skin incision, then after 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes from the start of anesthesia.
  millimeter mercury
Mean heart rate (HR) | basal, 5 minutes after the onsite of infiltration, 3 minutes after the onsite of skin incision, then after 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes from the start of anesthesia.
  beats per minute
Inhalational isoflurane concentration | intraoperative: at 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes from the start of anesthesia induction.
  percent
The number of hypertensive episodes | intraoperative
  defined as more than 25% rise of MBP than the basal, provided as total number
The number of tachycardic episodes | intraoperative
  defined as more than 25% rise of HR than the basal, provided as total number
Ephedrine consumption | intraoperative
  milligram
The total amount of fluid utilization. | intraoperative
  milliliter
Visual analog score | postoperative at 1,4,8,12,16, 20, 24 hours
  scale (0-10), 0= no pain
the time to first analgesic request | postoperative for 24 hours
  minutes
Opioid request episodes | postoperative for 24 hours
  number
Ambulation time | postoperative, the first test after 12 hours, then every 8 hours, up to 72 hours.
  hours to the time of first standing alone after the operation.
Hospital stay | postoperative, till the time of signed discharge order. up to 10 days
  days until the discharge time with the ability to walk, eat, controlled pain.
the Incidence of wound complications. | postoperative till 2 weeks
  infection, dehiscence, seroma, hematoma, bleeding
Surgeon satisfaction with the operative filed | within 2 hours from the end of operation
  score (0-10), 10 is the best
Patient satisfaction with analgesia | 24 hours after the end of surgery
  score (0-10), 10 is the best
Urine output | intraoperative
  milliliter

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital and Delta Hospital, Al Mansurah, Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: no limits
Access Criteria: e mail: alaa_mazy@yahoo.com